CLINICAL TRIAL: NCT03962829
Title: The Effect of Oral Administration of Meta-chlorophenylpiperazine (mCPP) on Cognitive Processes, Appetite, and Related Neural Responses in Healthy Lean and Obese Participants
Brief Title: Effect of mCPP on Cognitive Control, Appetite, and Neural Responses
Acronym: mCPP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: due to the Covid 19 pandemic
Sponsor: University of Birmingham (Other)
Collaborators: University Hospital Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: RG_16_214
Record Dates: First submitted 2019-05-22; First posted 2019-05-24 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Eating Behavior; Obesity
MeSH Terms: conditions — Feeding Behavior; Obesity | interventions — 1-(3-chlorophenyl)piperazine

STUDY DESIGN:
Intervention Model Description: counter-balanced, double-blind, placebo-controlled, crossover, within-subject design
Who Masked: Participant, Care Provider, Investigator
Masking Description: The research will be double blind; both placebo and mCPP will be presented in an identical capsule, therefore the participants and researchers do not know which treatment the participants will receive. A qualified pharmacist will follow standard operating procedures to encase the pharmacy prepared medications in a gelatine capsule in order to match the size and the appearance of the placebo. An independent researcher will prepare counterbalanced randomisation in advance.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo condition (Placebo Comparator): Participants receive placebo capsule
  Interventions: Drug: Placebo oral tablet
- mCPP condition (Active Comparator): Participants receive active (mCPP) capsule
  Interventions: Drug: mCPP

INTERVENTIONS:
Drug: mCPP — Healthy participants administrate one capsule of mCPP (30mg)
  Other Names: meta-chlorophenylpiperazine
  Arms: mCPP condition
Drug: Placebo oral tablet — Healthy participants administrate one capsule of placebo (containing lactose)
  Arms: Placebo condition

SUMMARY:
Previous studies have reported that the 5-HT2C receptor agonist meta-chlorophenylpiperazine (mCPP) decreases appetite and food intake in humans1-3. 5-HT2C receptor activation inhibits dopamine and norepinephrine release in the brain4, and has also been linked to diabetes5. The specificity of the effect of mCPP on human appetite is unclear, as previous studies also reported an increase in nausea1,3. The drug has also been reported to increase anxiety and cause panic attacks when given in a bolus dose intravenously6. Previous findings in our laboratory showed that mCPP reduced appetite, increased satiety in women and enhanced memory in the P1vital® Oxford Emotional Test Battery3. Following up on these results a food intake and fMRI study was performed, in which it was observed that mCPP decreased intake of a palatable snack (hedonic eating) and dlPFC and insula BOLD responses to food pictures. Additionally it increased memory and food value responses in brain after mCPP administration (Thomas et al submitted).

It is well established that eating behaviour is affected by metabolic signals (e.g. insulin, ghrelin, serotonin) and is also modulated via food reward processes7. More recently it has been proposed that eating is also modulated via higher cognitive processes such as inhibitory control, attention, and memory. However, in humans, eating behaviour seems to be a more complex process, which involves habits, long-term goals and social interaction. Thus, cognitive processes appear to play an important role in food consumption. In the proposed study the researchers investigate the effect of administering mCPP, on eating, and on metabolic, reward and cognitive processes and the potential interplay between these functions.

DETAILED DESCRIPTION:
The prevalence of overweight and obesity has increased rapidly in less than half a century. It is assumed that this development is due to interplay between behavioural, environmental and genetic factors. This increase in weight is associated with multiple-medical conditions, e.g. increased depression, and chronicle health conditions, like heart disease, cancer, and type 2 diabetes, and is associated with high health care costs. The UK has one of the highest rates of obesity in Europe, with 20% of the population defined as obese and over 50% defined as overweight. However treatment options for weight loss, and especially long-term weight maintenance are still limited. The development of safe and effective therapeutics is therefore imperative. An effective way to help weight loss, as part of a comprehensive program, is to prescribe drug treatments designed to reduce food consumption. However, at present, drug treatments for obesity are very limited.

mCPP appears to reduce food intake, and appetite in lean people. However it also seems to effect cognitive processes. Basic research to understand the interplay between these processes in relation to drug effects on appetite are of great interest because it can provide important insight into new development novel treatments for obesity. The investigators propose to test a model outlining that metabolic signals may reduce food intake by interfering with cognitive processes that underpin appetite.

It has been agreed upon that eating behaviour is affected by metabolic signals, e.g. serotonin, insulin and ghrelin, and influenced by food reward processes (Berthoud 2011). But the idea that these mechanisms are modulated via higher cognitive processes such as inhibitory control, attention, and memory is a relatively new domain to be explored. In humans, eating behaviour seems to be a more complex system; which also involves habits, long-term goals, and social interaction. Cognitive processes appear to play an important role in food consumption. Previous studies reported the anorectic effect of the drugs meta-chloriphenylpiperazine (mCPP), a 5-HT2C receptor agonist. Additionally mCPP has been shown to reduce appetite, increase satiety, and enhance memory for emotional material (word recall) and recognition memory (Thomas et al 2015). Preliminary results suggest that mCPP decreased intake of palatable snacks (hedonic eating) and when viewing food pictures appetite and reward related neural responses appear to be modulated by mCPP administration (Thomas et al in preparation). However the interaction between the drugs, neural responses and behaviour are still not known, and the effects of overweight on these responses is a very interesting question in relation to anti-obesity drug development.

In the proposed study the researchers want to investigate the effect of oral administrating mCPP, on neural responses and networks in relation to food reward, cognitive control and working memory and its impact on subsequent snack consumption, food and emotion related memory, and mood and appetite ratings, and additionally the interplay between all these processes in both lean and obese individuals. Participants will get an mCPP dose (30mg) and a placebo on different occasion, where after the neural activation (with fMRI) in response to food stimuli is assesed, inhibition tasks, and memory tests. This will be related to eating behaviour, memory performance, and mood and appetite ratings.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female subjects
* Age 18-65 years at start of the study
* Body Mass Index (BMI) between 18 and 25 kg/m2 for the lean group and between 30 and 40 kg/m2 for the obese group
* Right-handedness (including left-handers could bias the results because of the laterality of brain functions)
* Ability to give informed consent
* Fluent English speaking
* Willingness to be informed about chance findings of pathology

Exclusion Criteria:

* Subjects who have a non-removable metal object in or at their body, such as, for example: Heart pace-maker, artificial heart valve, metal prosthesis, implants or splinters, non-removable dental braces
* Tattoos, that are older than 15 years
* Claustrophobia
* Limited temperature perception and/or increased sensitivity to warming of the body
* Pathological hearing ability or an increased sensitivity to loud noises
* Lack of ability to give informed consent
* Operation less than three months ago
* Simultaneous participation in other studies that involve drugs intake or blood spending
* Acute illness or infection during the last 4 weeks
* Cardiovascular disorders (e.g., hypertrophic cardiomyopathy, long QT syndrome)
* Moderate or severe head injury
* Eating disorders
* No metabolic (e.g. metabolic disorder, diabetes, insulin resistance), psychological (e.g. depression) or neurological (e.g. epilepsy, headache disorder, multiple sclerosis, traumatic brain injuries) diseases or medication in relation to these diseases.
* Intake of any medication that can interfere with the drug or measurements.
* Current weight loss regimens, or more then 5kg weight loss in the last 3 months
* Smoking
* Current pregnancy or breastfeeding
* Current or past history of drug or alcohol dependency - alcohol consumption exceeding 12 units a week
* Food allergies (e.g. peanut allergy lactose and gluten intolerance) or vegetarian/vegan diet
* Disliking the study lunch

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — We aim to recruit 50% male and 50% female particpants
Enrollment: 32 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2020-03-20 (Actual)

PRIMARY OUTCOMES:
fMRI brain response during food reward processes | 21 min
  Brain responses for food stimuli compared to non-food stimuli. The researchers will measure this by showing subjects food and non-food images while preforming and fMRI-scan and subtract activity during non-food images from the activity pattern when looking at food images.

SECONDARY OUTCOMES:
fMRI brain response during inhibition processes | 20 min
  Neural activation during delay discounting paradigm for both food and monetary reward choices
Emotional categorisation | 10 min
  Accuracy of category and reaction time will be measured for dislike or like words
Emotional recall part 1 | 4 min
  Recall words of liked and disliked words will be recorded in ECAT
Emotional recall part 1 | 10 min
  Accuracy of previous exposed or not exposed words will be measured
Pasta intake | 20 min
  Amount (kcal and gram) of pasta eaten will be measured
Cookies intake | 10 min
  Amount (kcal and gram) of cookies eaten will be measured
fMRI neural network | 10 min
  Functional connectivity during resting state
VPA | 20 min
  Verbal pair association tasks, correct amount of word pairs remembered
N-back | 10 min
  N-back tasks, measure of working memory and working memory capacity

CONTACTS AND LOCATIONS:
Overall Officials: Maartje Spetter, PhD, Principal Investigator — University fo Birmingham
Locations (1):
- University of Birmingham School of Psychology, Birmingham, Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The study protocol and data will be shared on Open Science Forum
Supporting Information: Study Protocol
Time Frame: The study protocol and data will become available after the last participant has finished the study.
Access Criteria: All researchers
URL: https://osf.io